CLINICAL TRIAL: NCT05081622
Title: Preventing Violence by Teachers in Primary Schools in Haiti: A Cluster Randomized Controlled Trial of Interaction Competencies With Children - for Teachers (ICC-T)
Brief Title: Preventing Violence by Teachers in Primary Schools in Haiti
Acronym: ICC-T_HAITI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bielefeld University (Other)
Collaborators: University of Konstanz (Other); P4H Global (Unknown)
Responsible Party: Principal Investigator, Tobias Hecker, PhD, Assistant Professor, Bielefeld University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ICC-T_CRCT_Haiti
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: Violence by Teachers
Keywords: school violence; teacher violence; teachers; intervention; students; primary schools

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICC-T (Experimental): 5 days with 9 hours of training for teachers. Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting
  Interventions: Behavioral: Interaction Competencies with Children - for Teachers (ICC-T)
- Monitoring condition (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Interaction Competencies with Children - for Teachers (ICC-T) — Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting.
  A one-day ICC-T refresher workshop aiming to refresh and re-emphasize the key aspects of the intervention is implemented about 6 to 12 months after the initial intervention.
  Arms: ICC-T

SUMMARY:
Violence has severe and long-lasting negative consequences for children's and adolescents' well-being and academic functioning, which can hinder communities' and societies' economic growth. According to the Human Development Index, Haiti is one of the least developed countries in the world and the least developed in the Western hemisphere. Although Haiti has officially signed international and national laws aiming to protect children, preliminary reports suggest high rates of violence against children at schools. In addition to a lack of adequate training and supervision of teachers and an underdeveloped education system, attitudes favoring violence against children as an effective and acceptable discipline method and the lack of access to alternative non-violent strategies are likely to contribute to teachers' ongoing use of violence against children.

Notwithstanding, no school-level interventions addressing these factors to reduce violence by teachers have been scientifically evaluated in Haiti so far.

Thus, the present study tests the effectiveness of the preventative intervention Interaction Competencies with Children - for Teachers (ICC-T) in primary schools in Haiti. Previous studies have provided initial evidence on the feasibility and effectiveness of ICC-T to reduce teacher violence in primary and secondary schools in Tanzania and secondary schools in Uganda. This study aims to provide first evidence for the effectiveness of ICC-T to reduce violence and to improve children's functioning (i.e. mental health, well-being, academic performance) in a cultural setting outside of Sub-Saharan Africa.

DETAILED DESCRIPTION:
The study is designed as a two-arm cluster randomized controlled trial with schools (clusters) as level of randomization. The study will be conducted in the Northern department of Haiti. Six schools in each of the 6 included communes will be randomly selected, resulting in a total number of 36 schools.

In each commune, three schools will be randomly allocated to the intervention group (that will receive the ICC-T intervention) and three schools to the control group (that will receive no intervention). At each school, 28 students (stratified by gender) in the 4th grade of primary School (between 9 and 11 years of age) and all teachers (at least 13) will be recruited. Thus, the final sample will comprise at least 1008 students and at least 468 teachers.

The study will have two data assessment points: baseline assessment prior to the intervention and follow-up assessment six to 12 months after the intervention. In addition, feasibility data will be assessed in the intervention group at the beginning and the end of the intervention. Primary outcome measures are student- and teacher-reported physical and emotional violence by teachers in the past week. Secondary outcome measures include teachers' attitudes towards violence against students, children's emotional and behavioral problems, quality of life, and cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (if underaged by parents & minors themselves)

Students: Enrollment in class 4 of primary school

Teachers: All teachers employed at the school

Schools:

* Public or community schools
* Mixed-gender schools
* Day schools
* At least 40 students in selected class/stream

Exclusion Criteria:

Students and teachers:

* Acute drug or alcohol intoxication
* Acute psychotic disorder

Schools:

• Previous training on violence prevention

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1064 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change of students' exposure to emotional and physical violence by teachers | The CTS will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 6-12 months after intervention)
  The Conflict Tactics Scale (CTS) will be used to assess students' self-reported experiences of emotional and physical violence by teachers at school in the past week. Higher scores indicate higher levels of violence that is used by teachers. We hypothesize a stronger reduction of exposure to violence in the intervention group compared to the control group.
Change of teachers' use of emotional and physical violence | The CTS will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 6-12 months after intervention)
  The Conflict Tactics Scale (CTS) will be used to assess teachers' use of emotional and physical violent discipline measures against students in the past week. Higher scores indicate higher levels of violence that is used by teachers. We hypothesize a stronger reduction of the use of violence in the intervention group compared to the control group.

SECONDARY OUTCOMES:
Change of teachers' positive attitudes towards emotional and physical violence | The adapted version of CTS will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 6-12 months after intervention)
  Teacher's attitudes towards emotional and physical violence will be assessed with an adapted version of the Conflict Tactic Scale (CTS). Higher scores indicate higher levels of positive attitudes towards violence. We hypothesize a stronger decrease of positive attitudes towards violence in the intervention group compared to the control group.
Change of student's mental health | The PSC-Y will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 6-12 months after intervention)
  The Pediatric Symptom Checklist - Youth Report (PSC-Y) will assess students' emotional and behavioral problems.
  Higher scores indicate higher levels of students' mental health problems. We hypothesize a stronger reduction of mental health problems in the intervention group compared to the control group.
Change of students' quality of life | The KIDSCREEN-10 will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 6-12 months after intervention)
  The KIDSCREEN-10 will assess students' quality of life. Higher scores indicate higher levels of students' quality of life.
  We hypothesize a stronger increase of quality of life in the intervention group compared to the control group.
Change of students' cognitive functioning | The app-based tasks will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 6-12 months after intervention)
  Four tasks from the tablet application Psych Lab 101 will be used to assess children's cognitive abilities including selective attention, working memory, interference control and impulsivity. Higher scores indicate higher levels of students' cognitive abilities. We hypothesize higher levels of cognitive functioning in the intervention group compared to the control group.

OTHER OUTCOMES:
Change of students' academic performance | he standardized achievement tests will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 6-12 months after intervention).
  Purpose-built tests will be used to assess students' numeracy and literacy skills. Higher scores indicate higher levels of students' academic skills. In addition, students' grades in the previous term's exams will be obtained from the school administration. A change in academic performance in the intervention group is hypothesized.
Change of Students' social competence | The Social Cognitive Map Technique - peer nomination will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 6-12 months after intervention).
  The Social Cognitive Map Technique will assess students' social competence through peer nominations. Higher scores indicate higher levels of students' social competence. We hypothesize a stronger increase of social competence in the intervention group compared to the control group.
Change of peer violence | The Multidimensional Peer Victimization Scale will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 6-12 months after intervention).
  The Multidimensional Peer Victimization Scale will be used assess students' experiences of violence by peers. Higher scores indicate higher levels of students' experiences of peer violence. We hypothesize a stronger decrease of peer violence in the intervention group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Anke Hoeffler, Prof. Dr., Principal Investigator — University of Konstanz
Locations (1):
- P4H Global, Cap-Haïtien, Haiti

IPD SHARING:
Plan to Share IPD: No